CLINICAL TRIAL: NCT03636828
Title: Gastric Emptying Time of a Rice-based Meal Using Serial Sonographic Assessment
Brief Title: Gastric Emptying Time of a Rice-based Meal
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kangbuk Samsung Hospital (Other)
Responsible Party: Principal Investigator, Taejong Song, Professor, Kangbuk Samsung Hospital
Other Study IDs: KBSMC2018-08-001
Record Dates: First submitted 2018-08-06; First posted 2018-08-17 (Actual); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Gastric Emptying

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: ultrasonographic measurement of gastric antral cross-sectional area — Each participant fasted for 10 hours and subjected to a baseline gastric ultrasound and serial sonographic gastric evaluations was performed every hour after 2 hours of the ingestion of a 420 g, 536 Kcal rice-based meal (bibimbap) until the stomach was completely empty.

SUMMARY:
Adequate preoperative fasting is critical in preventing pulmonary aspiration of gastric content. Ultrasonography is considering as a useful test assessing the volume of gastric contents, but the emptying time of a rice-based meal (Asian foods) in healthy populations was not clear. The objective of this study was to investigate the minimum fasting time required for adequate gastric emptying after the ingestion of a rice-based meal.

DETAILED DESCRIPTION:
Aspiration of gastric contents into the lungs in surgical patients is a rare, but serious adverse event. Because a proper preoperative fasting is mandatory before anesthesia to prevent this severe complication, patients undergoing elective surgery have traditionally asked to fast overnight to ensure that their stomachs are empty. However, it is difficult and uncomfortable for patients not to eat or drink, particularly for those scheduled for surgery later in the day. Fasting may lead to thirst, hunger, anxiety, and tiredness, along with the potential for hypoglycemia and dehydration. Moreover, prolonged preoperative starvation triggers a metabolic response that precipitates gluconeogenesis and increases the organic response to trauma [7,8] and leads to delayed recovery after surgery. Avoiding inordinate fasting before surgery markedly reduces postoperative insulin resistance which has beneficial effects on postoperative glucose and protein metabolism.

Current guidelines by the American Society of Anesthesiologists (ASA) recommend a minimum of 6 hours after a light meal (toast and clear fluid) and 8 hours if the meal includes fried or fatty foods. In the era of evidence-based medicine, however, these fasting recommendations to keep a patient in preoperative fasting of 6-8 hours after the intake of solid meal are derived from survey opinions solicited from 470 active members of the ASA membership despite insufficient literature.

Recent studies have shown that real-time ultrasonography can provide reliable information about the nature (clear fluid, solid, or none) and volume of gastric content, being a non-invasive, inexpensive and safe method. The ultrasonographic measurement of antral cross-sectional area (CSA) is used for the assessment of gastric emptying in diabetic or dyspeptic patients and clinical investigations in obstetrical anesthesia. Thus, we designed this study to evaluate scientifically the gastric emptying time of solid meal using serial sonographic assessment in healthy volunteers. (Especially, there was no study to evaluate the gastric emptying time of a rice-based meal.) The objective of this study was to confirm or confront the minimum fasting time required for adequate gastric emptying for a rice-based meal (Asian foods), according to the suggestion of current guideline.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years old
* body mass index between 18.5 and 29.9 kg/m2

Exclusion Criteria:

* history of gastrointestinal disease such as history of surgery of upper abdomen, hiatal hernia and gastroesophageal reflux,
* diabetes mellitus
* chronic kidney disease
* pregnancy

Ages: 18 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: Study population is 10 healthy volunteers.
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2018-10-15 (Actual); Primary Completion 2018-12-27 (Estimated); Study Completion 2018-12-27 (Estimated)

PRIMARY OUTCOMES:
ultrasonographic measurement of gastric antral cross-sectional area (CSA) | 2 hours after the ingestion of a sold meal
ultrasonographic measurement of gastric antral cross-sectional area (CSA) | 3 hours after the ingestion of a sold meal
ultrasonographic measurement of gastric antral cross-sectional area (CSA) | 4 hours after the ingestion of a sold meal
ultrasonographic measurement of gastric antral cross-sectional area (CSA) | 5 hours after the ingestion of a sold meal
ultrasonographic measurement of gastric antral cross-sectional area (CSA) | 6 hours after the ingestion of a sold meal
ultrasonographic measurement of gastric antral cross-sectional area (CSA) | 7 hours after the ingestion of a sold meal
ultrasonographic measurement of gastric antral cross-sectional area (CSA) | 8 hours after the ingestion of a sold meal

CONTACTS AND LOCATIONS:
Overall Officials: Taejong Song, MD, PhD, Principal Investigator — Kangbuk Samsung Hosptial
Locations (1):
- Kangbuk Samsung Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No